CLINICAL TRIAL: NCT01076504
Title: A Phase II Trial of Amrubicin and Carboplatin With Pegfilgrastim in Patients With Extensive-Stage Small Cell Lung Cancer
Brief Title: A Trial of Amrubicin and Carboplatin With Pegfilgrastim in Patients With Extensive-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI LUN 199
Record Dates: First submitted 2009-12-08; First posted 2010-02-26 (Estimated); Results first posted 2015-12-10 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-04

CONDITIONS: Extensive-Stage Small Cell Lung Cancer
Keywords: SCLC; Amrubicin; Carboplatin; Pegfilgrastim; Neulasta
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — amrubicin; Carboplatin; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Amrubicin/Carboplatin with Pegfilgrastim (Experimental): Systemic therapy
  Interventions: Drug: Amrubicin; Drug: Carboplatin; Drug: Pegfilgrastim

INTERVENTIONS:
Drug: Amrubicin — 30 mg/m2 IV on Days 1-3 of each 3-week treatment cycle
  Other Names: SM-5887
Drug: Carboplatin — AUC=5 IV, Day 1 of each 3-week treatment cycle
  Other Names: cis-Diammine; Paraplatin; Paraplatin-AQ
Drug: Pegfilgrastim — 6 mg SQ on Day 4 of each 3 week treatment cycle
  Other Names: Neulasta

SUMMARY:
This proposed trial will investigate the combination of amrubicin and carboplatin in the first-line treatment of patients with extensive-stage small cell lung cancer (ES- SCLC). Since myelosuppression is the most common toxicity produced by this drug combination, pegfilgrastim will be administered with each treatment cycle. This trial will be the first clinical trial to evaluate a combination of amrubicin and carboplatin in the first-line treatment of ES SCLC in a U.S. population.

ELIGIBILITY:
Inclusion Criteria:

1. Cytologically and/or histologically confirmed small-cell lung cancer with extensive stage disease.
2. Measurable or evaluable disease per RECIST criteria version 1.1.
3. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0-1.
4. Left ventricular ejection fraction (LVEF) ≥50% by echocardiogram (ECHO) or multiple gated acquisition scan (MUGA).
5. QTc interval of ≤450 msec. on ECG.
6. Adequate organ function, including the following:

   * ANC ≥1500 cells/micro liter
   * Platelet count ≥100,000 cells/micro liter
   * Hemoglobin ≥9 g/dL
   * Total bilirubin ≤1.5 x ULN; AST/ALT ≤2.5 x ULN, (except if due to hepatic metastases, then ≤5 x ULN)
   * Serum creatinine ≤1.5 x ULN
7. Patients must be able to receive growth factors (G-CSF).
8. Women of childbearing potential must have a negative serum or urine pregnancy test performed ≤ 7 days prior to start of treatment. Women of childbearing potential or men with partners of childbearing potential must use effective birth control measures during treatment. If a woman becomes pregnant or suspects she is pregnant while participating in this study, she must agree to inform her treating physician immediately.
9. Patients ≥18 years of age.
10. Patients must be accessible for treatment and follow-up.
11. Patients must be able to understand the investigational nature of this study and give written informed consent prior to study entry.

Exclusion Criteria:

1. Previous treatment for limited-stage SCLC.
2. Previous chemotherapy or radiation therapy for SCLC (unless radiation was administered for brain metastases).
3. Active brain metastases. Patients with treated brain metastases are eligible, if (1) radiation therapy was completed ≥ 21 days prior to first dose of amrubicin; (2) follow-up scan shows no disease progression; an absence of neurologic symptoms and (3) patient does not require steroids.
4. Mixed small cell/non-small cell tumors or other neuroendocrine lung cancers.
5. Women who are pregnant or breastfeeding.
6. Suspected, diffuse idiopathic interstitial lung disease or pulmonary fibrosis.
7. Patients with New York Heart Association (NYHA) class II or greater congestive heart failure (CHF).
8. Any of the following ≤6 months prior to starting study treatment:

   * myocardial infarction;
   * severe unstable angina;
   * ongoing cardiac dysrhythmia.
9. Family history of idiopathic cardiomyopathy or uncontrolled heart arrhythmia.
10. Treatment for other invasive cancers during the previous 5 years, or the presence of any active invasive cancer of any type (with the exception of non-melanoma skin cancers).
11. Uncontrolled hypertension (i.e., blood pressure >150/90 mmHg that cannot be controlled with standard anti-hypertensive agents).
12. Major surgical procedure or significant traumatic injury ≤ 28 days of study initiation.
13. History of seropositive HIV or patients who are receiving immunosuppressive medications that would in the opinion of the investigator increase the risk of the serious neutropenic complications.
14. Concurrent severe, intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements.
15. Any condition that would prevent patient comprehension of the nature of, and risk associated with, the study.
16. Use of any non-approved or investigational agent ≤30 days prior to administration of the first dose of study drug. Patients may not receive any other investigational or anti-cancer treatments while participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2009-12; Primary Completion 2012-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R Spigel, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (20):
- United States (20):
  - Northeast Arkansas Clinic, Jonesboro, Arkansas
  - Florida Cancer Specialists, Fort Myers, Florida
  - Watson Clinic Center for Cancer Care and Research, Lakeland, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Medical Oncology Associates of Augusta, Augusta, Georgia
  - Baptist Hospital East, Louisville, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Hematology Oncology Clinic, LLP, Baton Rouge, Louisiana
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - National Capital Clinical Research Consortium, Bethesda, Maryland
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Research Medical Center, Kansas City, Missouri
  - Nebraska Methodist Cancer Center, Omaha, Nebraska
  - Oncology Hematology Care, Cincinnati, Ohio
  - South Carolina Oncology Associates, PA, Columbia, South Carolina
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Family Cancer Center, Collierville, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Peninsula Cancer Institute, Newport News, Virginia
  - Virginia Cancer Institute, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 81 patients were enrolled but 1 patient was hospitalized prior to receiving any protocol treatment and was never treated. 80 patients included in the analysis
Period: Overall Study
Arm/Group | Amrubicin/Carboplatin With Pegfilgrastim
Started | 80
Completed | 0 (Patients remained on study until disease progression or withdrawal for any other reason)
Not Completed | 80

BASELINE CHARACTERISTICS:
Population: 81 patients were enrolled but 1 patient was hospitalized prior to receiving any protocol treatment and was never treated. 80 patients included in the analysis
Arm/Group | Amrubicin/Carboplatin With Pegfilgrastim
Number analyzed (Participants) | 80
Age, Continuous [Median (Full Range); unit: years] | 65 [45 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 36
Region of Enrollment [Number; unit: participants]
  United States | 80

OUTCOME MEASURES:

1. Primary Outcome: 1-year Survival
Description: Percentage of patients still alive one year after their first treatment
Time Frame: 12 months
Population: All enrolled and treated patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Amrubicin/Carboplatin With Pegfilgrastim
Number analyzed (Participants) | 80
percentage of participants | 38 [25 to 50]

2. Secondary Outcome: Objective Response Rate
Description: The Percentage of Patients Who Experience an Objective Benefit From Treatment. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI or CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Objective Response (OR) = CR + PR.
Time Frame: 36 months
Population: Includes all patients who were treated and evaluated for response (74 patients - 6 were deemed not evaluable)
Measure: Number; unit: percentage of evaluable participants
Arm/Group | Amrubicin/Carboplatin With Pegfilgrastim
Number analyzed (Participants) | 74
percentage of evaluable participants | 80

3. Secondary Outcome: Time to Progression
Description: Time to progression will be defined as the time from first treatment until objective tumor progression (PD). Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 36 months
Population: Includes all enrolled and treated patients
Measure: Median (Full Range); unit: weeks
Arm/Group | Amrubicin/Carboplatin With Pegfilgrastim
Number analyzed (Participants) | 80
weeks | 23 [1.4 to 104.4]

4. Secondary Outcome: Overall Survival
Description: The Length of Time, in Months, That Patients Were Alive From Their First Date of Protocol Treatment Until Death
Time Frame: 84 months
Population: All enrolled and treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Amrubicin/Carboplatin With Pegfilgrastim
Number analyzed (Participants) | 80
months | 10.3 [8.5 to 13]

5. Secondary Outcome: Toxicity/Safety
Description: Grade 3/4 toxicities
Time Frame: 36 months
Population: All enrolled and treated patients
Measure: Number; unit: participants
Arm/Group | Amrubicin/Carboplatin With Pegfilgrastim
Number analyzed (Participants) | 80
participants
  Anemia | 22
  Leukopenia | 30
  Thrombocytopenia | 36
  Neutropenia | 29
  Febrile neutropenia | 10
  Hypokalemia | 14
  Fatigue | 11
  Dehydration | 8
  Infection | 11
  Hyponatremia | 10
  Nausea | 8
  Vomiting | 6
  Hyperglycemia | 3
  Muscle weakness | 4
  Thrombosis/embolism | 3

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Amrubicin/Carboplatin With Pegfilgrastim
Serious Adverse Events (participants affected / at risk) | 0/80
Other Adverse Events (participants affected / at risk) | 80/80
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Amrubicin/Carboplatin With Pegfilgrastim (N=80)
Allergic reaction (Immune system disorders) | 80
Anemia (Blood and lymphatic system disorders) | 80
ANOREXIA (Metabolism and nutrition disorders) | 80
CONSTIPATION (Gastrointestinal disorders) | 80
DEHYDRATION (Metabolism and nutrition disorders) | 80
DIARRHEA (Gastrointestinal disorders) | 80
Dizziness (Nervous system disorders) | 80
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 80
FATIGUE (General disorders) | 80
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 80
Fever (General disorders) | 80
Gastrointestinal disorders - Other, stomatitis (Gastrointestinal disorders) | 80
HYPOKALEMIA (Metabolism and nutrition disorders) | 80
Infections and infestations - Other, pneumonia (Infections and infestations) | 80
MYALGIA (Musculoskeletal and connective tissue disorders) | 80
NAUSEA (Gastrointestinal disorders) | 80
Neutrophil count decreased (Investigations) | 80
PAIN (General disorders) | 80
Platelet count decreased (Investigations) | 80
VOMITING (Gastrointestinal disorders) | 80
Weight loss (Investigations) | 80
White blood cell decreased (Investigations) | 80
Alopecia (Skin and subcutaneous tissue disorders) | 35
generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 31
Hypoalbuminemia (Metabolism and nutrition disorders) | 29
hyperglycemia (Metabolism and nutrition disorders) | 26
Hyponatremia (Metabolism and nutrition disorders) | 25
Alkaline phosphatase increased (Investigations) | 23
Cough (Respiratory, thoracic and mediastinal disorders) | 20
Insomnia (Psychiatric disorders) | 18
Hypocalcemia (Metabolism and nutrition disorders) | 17
edema limbs (General disorders) | 16
Hypotension (Vascular disorders) | 16
Blood bilirubin increased (Investigations) | 15
Investigations - Other, blood protein decreased (Investigations) | 15
Investigations - Other, blood urea nitrogen increased (Investigations) | 14
Investigations - Other, creatinine decreased (Investigations) | 14
Cardiac disorders - Other, tachycardia (Cardiac disorders) | 13
Depression (Psychiatric disorders) | 13
Investigations - Other, blood chloride decreased (Investigations) | 13
Hypomagnesemia (Metabolism and nutrition disorders) | 12
Investigations - Other, blood urea nitrogen decreased (Investigations) | 12
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 12
Dysgeusia (Nervous system disorders) | 11
Hyperkalemia (Metabolism and nutrition disorders) | 11
Investigations - Other, blood bicarbonate decreased (Investigations) | 11
Rash (Skin and subcutaneous tissue disorders) | 11
Skin and subcutaneous tissue disorders - Other, erythema (Skin and subcutaneous tissue disorders) | 11
abdominal pain (Gastrointestinal disorders) | 10
Anxiety (Psychiatric disorders) | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 10
Mucositis (Gastrointestinal disorders) | 10
Investigations - Other, blood bicarbonate increased (Investigations) | 9
Investigations - Other, blood chloride increased (Investigations) | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9
Dyspepsia (Gastrointestinal disorders) | 8
Chills (General disorders) | 7
confusion (Psychiatric disorders) | 7
Creatinine increased (Investigations) | 7
Fall (Injury, poisoning and procedural complications) | 7
Gastroesophageal reflux disease (Gastrointestinal disorders) | 7
Urinary Tract Infection (Infections and infestations) | 7
Bruising (Injury, poisoning and procedural complications) | 6
Hypertension (Vascular disorders) | 6
Lymphocyte count decreased (Investigations) | 6
Malaise (General disorders) | 6
Peripheral sensory neuropathy (Nervous system disorders) | 6
Thromboembolic event (Vascular disorders) | 6
Tremor (Nervous system disorders) | 6
Alanine aminotransferase increased (Investigations) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 5
Dysphagia (Gastrointestinal disorders) | 5
Headache (Nervous system disorders) | 5
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 5
Infections and infestations - Other, oral infection (Infections and infestations) | 5
Infections and infestations - Other, unspecified (Infections and infestations) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Proteinuria (Renal and urinary disorders) | 5
Somnolence (Nervous system disorders) | 5
flushing (Vascular disorders) | 4
Hypernatremia (Metabolism and nutrition disorders) | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4
Psychiatric disorders - Other, change in mental status (Psychiatric disorders) | 4
Respiratory, thoracic and mediastinal disorders - Other, decreased breath sounds (Respiratory, thoracic and mediastinal disorders) | 4
Sinusitis (Infections and infestations) | 4
Skin and subcutaneous tissue disorders - Other, decreased turgor (Skin and subcutaneous tissue disorders) | 4
Syncope (Nervous system disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 but =180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites